CLINICAL TRIAL: NCT00928798
Title: Topical Rapamycin to Treat Fibrofolliculomas in Birt-Hogg-Dubé Syndrome
Brief Title: Topical Rapamycin for Fibrofolliculomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Myrovlytis Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 09-2-058
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Birt-Hogg-Dubé Syndrome
MeSH Terms: conditions — Birt-Hogg-Dube Syndrome | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- rapamycin (Experimental): one facial side rapamycin and one facial side placebo
  Interventions: Drug: Rapamycin; Drug: placebo

INTERVENTIONS:
Drug: Rapamycin — Application of rapamycin 1 mg/ml oral solution to one predefined skin area on one facial half, twice daily 0,25 ml, during 6 months. The other facial half will be similarly treated with a placebo.
  Other Names: Rapamune; Sirolimus
Drug: placebo — Application of placebo to one predefined skin area on one facial half, during 6 months. The other facial half will be similarly treated with rapamycin 1 mg/ml oral solution

SUMMARY:
The purpose of the study is to determine whether topical application of rapamycin can lead to reduction in size and/or number of fibrofolliculomas in BHD patients and may prevent the growth of new ones. Secondary we evaluate rapamycin safety, formula acceptance and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years.
* At least 10 facial fibrofolliculomas, histologically confirmed.
* Entered in a screening program and free of malignancy as determined during screening (already had a baseline MRI or CT-scan).
* Being able to understand instructions.
* Mutation status must be known.
* For females: not pregnant and willing to use both oral and barrier contraceptives during the treatment period.

Exclusion Criteria:

* Not capable of informed consent.
* Age under 18 years.
* Pregnancy or failure to comply with contraceptive measures.
* Proven or suspected malignancy of skin or other organs.
* No histological confirmation.
* Skin lesions other than fibrofolliculoma that might worsen under sirolimus such as active infections.
* Not able to comprehend instructions.
* No proven mutation.
* Less than 10 fibrofolliculomas.
* Planned facial surgery in the treatment period.
* Concomitant disease requiring systemic immunosuppressive treatment
* Concomitant disease requiring facial topical immunosuppressive treatment or facial topical drugs that interfere with rapamycin during trail period or in the 30 days before start trial.
* Tendency to form keloids or hypertrophic scars.
* Drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Significant regression of lesions (reduction of fibrofolliculoma size and count) in the treated area. | 3 and 6 months

SECONDARY OUTCOMES:
Side effects | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurice van Steensel, Dr., Principal Investigator — Department of Dermatology
Locations (2):
- Netherlands (2):
  - VU Medical Centre Amsterdam, Amsterdam
  - Maastricht University Medical Centre, Maastricht

REFERENCES:
- [Derived] Gijezen LM, Vernooij M, Martens H, Oduber CE, Henquet CJ, Starink TM, Prins MH, Menko FH, Nelemans PJ, van Steensel MA. Topical rapamycin as a treatment for fibrofolliculomas in Birt-Hogg-Dube syndrome: a double-blind placebo-controlled randomized split-face trial. PLoS One. 2014 Jun 9;9(6):e99071. doi: 10.1371/journal.pone.0099071. eCollection 2014. PMID 24910976